CLINICAL TRIAL: NCT02173496
Title: Evaluation of Multiple Assessment Modalities for the Detection and Characterisation of the Preclinical, Pre-symptomatic Stage of Neovascular Age-related Macular Degeneration
Brief Title: Colour Contrast Sensitivity for the Early Detection of Wet Age-related Macular Degereration (CEDAR)
Acronym: CEDAR
Status: Completed | Type: Observational
Sponsor: Aston University (Other)
Collaborators: The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CEDAR001; 14/WM/0035 (Other: Solihull NRES Ethics Committee, UK)
Record Dates: First submitted 2014-03-20; First posted 2014-06-25 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Age Related Macular Degeneration
Keywords: Wet age-related macular degeneration; Assessment modalities for preclinical, pre-symptomatic ARMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colour contrast sensitivity: Colour contrast sensitivity
  Interventions: Other: Colour Contrast Sensitivity

INTERVENTIONS:
Other: Colour Contrast Sensitivity — Reading of numbers or letters from a monitor

SUMMARY:
Neovascular or wet age-related macular degeneration (ARMD) is a retinal disease and is the leading cause of sight loss in the over 50s; it constitutes a major public health problem which will have an increasingly large impact as the population ages, because sight loss has been associated with loss of independence, depression, social isolation, and falls.

Recent advances in medicine, and in particular the approval on behalf of the National Institute for Health and Clinical Excellence (NICE) for use of ranibizumab (Lucentis) in wet ARMD, have allowed this condition to be treated; however success is more likely when treatments occur at a very early stage.

Unfortunately the early stages of wet ARMD do not cause symptoms and most cases are diagnosed when irreversible retinal damage has already occurred.

In all stages of ARMD, even when no symptoms are present and non-invasive techniques currently used in routine clinical practice are not sufficiently sensitive to identify abnormalities, retinal function and possibly anatomy are abnormal.

This study will evaluate techniques that may be useful in flagging subjects with the "preclinical" stages of the disease. This may allow early preventative measures to be taken, in order to stop altogether the onset of blindness.

The study will focus mainly on colour contrast sensitivity, a simple but highly sensitive technique to assess retinal function, to establish if people with wet ARMD can be identified before symptoms develop. Other assessment modalities, evaluating either structure or function of the retina, will also be employed in selected individuals to establish if they may be used in the routine clinic; however it is already known that these modalities are not suitable for all individuals, as they are more demanding time-wise and concentration-wise, and therefore not universally suitable.

DETAILED DESCRIPTION:
Neovascular age-related macular degeneration (nARMD), which by definition affects the over 50s, accounts for more than 50% of visual impairment certifications in the United Kingdom1 and a recent study2 estimates the prevalence in the UK at 1.2% in individuals aged 50 or more, 2.5% in those over 65, and 6.3% in those aged 80 or more. Neovascular ARMD is therefore likely to become a much more significant issue as the population ages, unless steps are taken now to find ways of limiting loss of vision: the same study2 suggests there are currently 263,000 cases of nARMD in the UK, but the number is set to increase by almost a third by the year 2020. Importantly, individuals with poor vision also have a higher frequency of falls and of depression compared to aged-matched people with normal vision, and are likely to live alone and have additional health problems3, 4. Therefore nARMD significantly impacts on quality of life, to a much greater extent than appreciated by many health professionals: a key study5 reported that even mild sight impairment results in a 17% decrease in quality of life, whereas moderate and severe sight impairment result in a 40% and 63% decrease in quality of life respectively. It should be noted that a 63% decrease in quality of life is comparable to that encountered with advanced prostatic cancer with uncontrollable pain or a severe stroke that leaves a person bedridden, incontinent and requiring constant nursing care5.

The advent of anti-VEGF therapy in nARMD and the approval of ranibizumab (Lucentis) in the UK by the National Institute for Clinical Excellence (NICE) has dramatically improved the prognosis of patients with nARMD: vision can frequently be maintained or even improved, particularly if early detection and treatment occur6-9. However it is currently difficult to detect and monitor nARMD in its early stages and most individuals typically present to the ophthalmologist only once a certain degree of irreversible damage has occurred. The hallmark of nARMD is a choroidal neovascular membrane (CNV) 1, 10, 11, although changes occur locally before a CNV develops, as follows:

1. Inflammatory mediators are released in the affected area and changes in metabolism develop12-15.
2. The retina affected by the insult gradually loses its function10-12, 14-18. It has yet to be established at which point of CNV development the surrounding retina has detectable functional and structural abnormalities, however a wealth of literature10-12, 14-19 suggests it starts when the patient is still asymptomatic and before currently available non-invasive imaging techniques are able to detect any abnormality. Many studies10, 12, 17, 18, 20 indicate that the above mentioned changes in metabolism determine abnormal function in the overlying photoreceptors/inner retina very early in the disease process, with some cone populations affected more than others18, 20, 21. The same studies suggest it is possible to detect this localised abnormal retinal function early with colour contrast sensitivity (CCS), especially in the blue-yellow (tritan) axis. The investigators therefore propose this technique can be utilised to identify people at risk of developing nARMD and those with the early, presymptomatic stage of the disease. The study will also evaluate other modalities which test either structure or function of the retina, to establish if any can be used for the early detection of nARMD.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years of age
* Unilateral wet ARMD

Exclusion Criteria:

* Bilateral wet ARMD
* Other retinal pathology
* High refractive error
* Not fluent in English
* Unable to give informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unilateral wet ARMD
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Capability of evaluated techniques detecting asymptomatic wet ARMD | 24 months

SECONDARY OUTCOMES:
Improve understanding of the disease process in wet ARMD | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Calcagni, MD, Principal Investigator — Aston University
Locations (1):
- Aston University, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No